CLINICAL TRIAL: NCT01540578
Title: OBSERVATIONAL: Replication Profiling as a Diagnostic Tool in B-cell Acute Lymphoblastic Leukemia (ALL)
Brief Title: Studying Biomarkers as a Diagnostic Tool in Samples From Younger Patients With B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B3; NCI-2012-00685 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-22; First posted 2012-02-29 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: B-cell Childhood Acute Lymphoblastic Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fresh and frozen bone marrow cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: Archived cell samples are analyzed for replication timing by flow cytometry, microarray, and single-cell fluorescence in situ hybridization (FISH) assays. Replication-timing results among cases and controls are also analyzed.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial is studying biomarkers as a diagnostic tool in samples from younger patients with B-cell acute lymphoblastic leukemia. Finding specific biomarkers may help improve the treatment of patients with B-cell acute lymphoblastic leukemia

DETAILED DESCRIPTION:
STUDY SUBTYPE: Ancillary/Correlative

OBSERVATIONAL STUDY MODEL: Case-only

TIME PERSPECTIVE: Retrospective

BIOSPECIMEN RETENTION: Samples with DNA

BIOSPECIMEN DESCRIPTION: Fresh and frozen bone marrow cells

STUDY POPULATION DESCRIPTION: Patients with B-cell acute lymphoblastic samples banked at the COG Cell Bank

SAMPLING METHOD: Non-probability sample

OBJECTIVES:

I. To determine whether we can identify individuals within a specific sub-group of pre-B acute lymphoblastic leukemia (ALL) patients that will eventually recur.

II. To identify replication-timing changes as a biomarker for further risk prediction.

III. To identify differences between patients of similar subtype, and choose candidate differences to analyze by methods that are compatible with frozen samples.

OUTLINE:

Archived cell samples are analyzed for replication timing by flow cytometry, microarray, and single-cell fluorescence in situ hybridization (FISH) assays. Replication-timing results among cases and controls are also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Frozen viable cell samples from patients with B-cell acute lymphoblastic (ALL) of any outcome from the Children's Oncology Group (COG) ALL Cell Bank (Part 1)
* Freshand frozen cell samples from patients with B-cell ALL with known outcomes from the COG ALL Cell Bank (Part 2) meeting 1 of the following criteria:

  * Samples from patients who experienced an early recurrence within 36 months of diagnosis (cases)
  * Samples from patients who remain in prolonged remission (controls)
* No samples meeting either of the following criteria:

  * Very-high-risk features

    * Philadelphia chromosome positive
    * Hypodiploid
    * MLL (11q23) rearranged
  * Known favorable risk factors

    * Hyperdiploid
    * t(12;21) (ETV6/RUNX1)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with B-cell acute lymphoblastic samples banked at the COG Cell Bank
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Replication-timing changes as a biomarker for further risk prediction by FISH | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: David Gilbert, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States